CLINICAL TRIAL: NCT02282605
Title: A Phase I/II Randomised, Double-blind, Placebo-controlled, Single Centre Study of the Nasal Decolonisation of Staphylococcus Aureus (SA) and the Safety and Tolerability of Two Concentrations of XF-73 Nasal Gel in Healthy Subjects.
Brief Title: Study of the Nasal Decolonisation of Staphylococcus Aureus (SA) and the Safety and Tolerability of XF-73 Nasal Gel in Healthy Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Destiny Pharma Plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XF-73B03
Record Dates: First submitted 2014-10-21; First posted 2014-11-04 (Estimated); Results first posted 2016-10-07 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-06

CONDITIONS: Staphylococcus Aureus Infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — chlorhexidine gluconate; Textiles

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- XF-73 2.0 mg/g nasal gel (Experimental): 0.3mL (nominal 300 microgram) XF-73 nasal gel will be applied to each naris, twice daily for two days. Each dose will be 0.3mL per naris/0.6mL per dose delivering 0.6mg XF-73 per naris/1.2mg XF-73 per dose. Prior to each morning dose, subjects will use chlorhexidine gluconate 2% body and face cloths.
  Interventions: Drug: XF-73 nasal gel; Other: Chlorhexidine gluconate 2% topical cloths
- XF-73 0.5 mg/g nasal gel (Experimental): 0.3mL (nominal 300 microgram) XF-73 nasal gel will be applied to each naris twice daily for two days. Each dose will be 0.3mL per naris/0.6mL per dose delivering 0.15mg XF-73 per naris/0.3mg XF-73 per dose. Prior to each morning dose, subjects will use chlorhexidine gluconate 2% body and face cloths.
  Interventions: Drug: XF-73 nasal gel; Other: Chlorhexidine gluconate 2% topical cloths
- Placebo nasal gel (Placebo Comparator): 0.3mL nasal gel will be applied to each naris twice daily for two days. Prior to each morning dose, subjects will use chlorhexidine gluconate 2% body and face cloths.
  Interventions: Drug: Placebo nasal gel; Other: Chlorhexidine gluconate 2% topical cloths

INTERVENTIONS:
Drug: XF-73 nasal gel
  Arms: XF-73 0.5 mg/g nasal gel; XF-73 2.0 mg/g nasal gel
Drug: Placebo nasal gel
  Arms: Placebo nasal gel
Other: Chlorhexidine gluconate 2% topical cloths

SUMMARY:
Study to determine the efficacy, safety and tolerability of two concentrations of XF-73 nasal gel in combination with body and face washing with chlorhexidine gluconate cloths in eradicating nasal carriage of Staphylococcus aureus.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy male or female subjects aged between 18 and 75 years.
2. Subjects confirmed to be persistent nasal SA carriers, defined by 3 separate, SA positive cultures from nasal swabs. Two positive cultures should be obtained at screening visits up to 12 weeks prior to inclusion and at least two weeks apart. The final confirmatory culture should be obtained from a nasal swab on the day of admission to the unit (day -1). Note: Dosing with XF-73 may commence before the result of the day -1 swab is obtained. If the result is negative, the subject should be withdrawn.
3. Subjects who are able and willing to provide written informed consent to participate in the study
4. Subjects who have a body mass index (BMI) ≥18.5 kg/m2 and ≤ 32kg/m2.
5. Subjects who agree not to take part in another clinical trial at any time during the study period.

Exclusion Criteria:

1. Female subjects who are or may be pregnant or who are lactating.
2. Subjects who have any acute or chronic illness or infection.
3. Subjects who have smoked within the 3 months prior to screening.
4. Subjects who are females of child-bearing potential, defined as being physiologically capable of becoming pregnant, UNLESS using one or more of the following acceptable methods of contraception; established use of oral, injected or implanted hormonal contraception, intrauterine Device (IUD or Coil AND barrier Method (condom or diaphragm or cervical/vault cap) plus spermicidal cream/gel. Contraceptive use should continue throughout the study and for 1 month following completion of the study.
5. Subjects who are fertile males, defined as all males physiologically capable of conceiving offspring, UNLESS the subject agrees to comply with acceptable contraception e.g. condom plus spermicidal cream/gel. Contraceptive use should continue throughout the study and for 3 months following completion of the study.
6. Subject with any open wound, lesion, inflammation, erythema or infection affecting the nostrils, nose, upper lip and area of skin close to the nose. This includes herpes simplex lesions and discoid lupus.
7. Subjects who have a currently symptomatic upper respiratory tract infection, nasopharyngitis, influenza or condition involving increase in nasal secretion such as seasonal or chronic, allergic rhinitis.
8. Subjects with a history of drug or alcohol abuse in the previous 12 months or who have a positive urine drug test for substances of abuse.
9. Subjects with a known clinically significant history of atopy or hypersensitivity to any drug or latex.
10. Subjects with a history of serious illness, cancer or psychiatric condition.
11. Subjects with known skin photosensitivity.
12. Subjects with a personal or family history of porphyria.
13. Subjects who have been treated with or have taken any prescribed or over-the-counter medication within the 14 days prior to admission, with the exception of hormonal contraceptives or hormone replacement therapy.
14. Subjects who have taken or used topical or systemic antibiotics within the month prior to screening.
15. Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or who have a positive result to the test for human immunodeficiency virus (HIV) antibodies
16. Subjects who have participated in a clinical trial within the last 3 months.
17. Subjects who have been exposed to XF-73 as part of a previous clinical trial.
18. Subjects with any clinically significant abnormality in vital signs or laboratory analyses at screening or at baseline, based on the opinion of the investigator.
19. Subjects with nasal polyps or significant anatomical nasal abnormality.
20. Subjects with a history of nasal surgery, including cauterization in the last 12 months.
21. Subjects with a history of multiple episodes [>3] of epistaxis within the last 12 months.
22. Subjects known to have dermal sensitivity to benzalkonium chloride or other quaternary ammonium disinfectants.
23. Subjects with in-situ nasal jewellery or open nasal piercings.
24. Subjects known to have dermal sensitivity to chlorhexidine gluconate (CHG).
25. Subjects with a history of abnormal bleeding, bruising, frequent nosebleeds or a diagnosis of von Willebrand disease.
26. Subjects who have or have had an autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Mr Hayter, BSc, Study Director — Destiny Pharma Plc
Locations (1):
- Quintiles Drug Research Unit, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Persistent nasal SA carriage was defined by 3 separate, SA positive cultures from nasal swabs. The protocol allowed for dosing to commence before the results of the final swab on day -1 were available. Dosing was thus commenced in 3 subjects in the XF-73 2.0mg/g group but was withdrawn as the day -1 SA results were negative.
Groups:
- XF-73 2.0 mg/g Nasal Gel: 0.3mL (nominal 300 microgram) XF-73 nasal gel will be applied to each naris, twice daily for two days. Each dose will be 0.3mL per naris/0.6mL per dose delivering 0.6mg XF-73 per naris/1.2mg XF-73 per dose. Prior to each morning dose, subjects will use chlorhexidine gluconate 2% body and face cloths.
  XF-73 nasal gel
  Chlorhexidine gluconate 2% topical cloths
- XF-73 0.5 mg/g Nasal Gel: 0.3mL (nominal 300 microgram) XF-73 nasal gel will be applied to each naris twice daily for two days. Each dose will be 0.3mL per naris/0.6mL per dose delivering 0.15mg XF-73 per naris/0.3mg XF-73 per dose. Prior to each morning dose, subjects will use chlorhexidine gluconate 2% body and face cloths.
  XF-73 nasal gel
  Chlorhexidine gluconate 2% topical cloths
- Placebo Nasal Gel: 0.3mL nasal gel will be applied to each naris twice daily for two days. Prior to each morning dose, subjects will use chlorhexidine gluconate 2% body and face cloths.
  Placebo nasal gel
  Chlorhexidine gluconate 2% topical cloths
Period: Overall Study
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel
Started | 27 | 12 | 24
Completed | 24 | 12 | 24
Not Completed | 3 | 0 | 0
Not completed — negative SA result on Day -1 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel | Total
Number analyzed (Participants) | 27 | 12 | 24 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (12.4) | 38.0 (12.8) | 39.0 (12.5) | 37.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 5 | 20
  Male | 15 | 9 | 19 | 43
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27 | 12 | 24 | 63

OUTCOME MEASURES:

1. Primary Outcome: Apparent Eradication of Nasal SA After the Last Dose of XF-73 Based on Semi-quantitative SA Scores From a Broth Enrichment Method.
Description: Anti-SA activity was assessed by the quantification of SA colonisation using the broth enriched (semi-quantitative culture) 0-6 point scale. Scores of negative and 0 were interpreted as absence of SA (Responder) and scores of 1 or greater were interpreted as presence of SA (Non-Responder).
Time Frame: The primary endpoint was 48 hours after the last dose (Day 4, 84 hours).
Population: Exploratory comparisons between active groups versus placebo of the number of Responder subjects were performed using a one-sided Fisher's exact test at 5% significance level.
Measure: Number; unit: participants
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel
Number analyzed (Participants) | 27 | 12 | 24
participants | 3 | 1 | 4
Statistical Analysis 1: Comparison: XF-73 2.0 mg/g Nasal Gel vs Placebo Nasal Gel; Test type: Superiority or Other; p = 0.792, Fisher Exact
Statistical Analysis 2: Comparison: XF-73 0.5 mg/g Nasal Gel vs Placebo Nasal Gel; Test type: Superiority or Other; p = 0.887, Fisher Exact

2. Secondary Outcome: Apparent Eradication of Nasal SA After the Last Dose of XF-73 Based on Semi-quantitative SA Scores From a Broth Enrichment Method.
Description: as for outcome 1
Time Frame: Time-points: Day 1(12 hours), Day 2 (24 hours), Day 3 (12 hours after last dose), Day 7 and Day 14.
Population: Exploratory comparisons between active groups versus placebo of the percentage of Responder subjects were performed using a one-sided Fisher's exact test at 5% significance level.
Measure: Number; unit: participants
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel
Number analyzed (Participants) | 27 | 12 | 24
participants
  Day 1 (12 hours) | 2 | 2 | 6
  Day 2 (24 hours) | 10 | 3 | 2
  Day 3 (12 hours after last dose) | 9 | 9 | 6
  Day 7 | 1 | 0 | 1
  Day 14 | 1 | 0 | 2
Statistical Analysis 1: Comparison: XF-73 0.5 mg/g Nasal Gel vs Placebo Nasal Gel; Test type: Superiority or Other; p = 0.0058, Fisher Exact — For timepoint Day 3 (12 hours after last dose)

3. Secondary Outcome: Time-point at Which Clearance Was First Observed From Nasal Swabs Based on Semi-quantitative Score
Description: The number of subjects with absence of SA from nasal swabs at the specified time-points..
Time Frame: Day 1 (12 h), Day 2 (24 h) , Day 3 (12 hours after last dose),Day 4 (48 hours after last dose)
Measure: Number; unit: participants
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel
Number analyzed (Participants) | 27 | 12 | 24
participants
  Day 1 (12 hours) | 1 | 2 | 5
  Day 2 (24 hours) | 8 | 2 | 1
  Day 3 (12 hours after last dose) | 4 | 5 | 4
  Day 4 (48 hours after last dose) | 0 | 0 | 1

4. Secondary Outcome: AUC of the Semi-quantitative SA Scores From Nasal Swabs
Description: Anti-SA activity was assessed by the quantification of SA colonisation using the broth enriched (semi-quantitative culture) 0-6 point scale. Mean changes from baseline (0h) to each timepoint (Day 1,12 h; Day 2, 24 h: Day 3, 48h; Day 4, 84h; Day 7, 144h; Day 14, 312h) were calculated by treatment for the semi-quantitative SA scores. The AUC of the semi-quantitative SA scores were calculated for the two-day treatment period (AUC Day1- Day2); through the two day treatment period and up to discharge (AUC Day 1- Day4); and over the two-day treatment period, discharge and follow-up (AUC Day1- Day14). AUC was calculated by means of a trapezoidal rule using a standard algorithm. A higher AUC is indicative of a higher bacterial growth.
Time Frame: 2 day treatment period; 2 day treatment period up to discharge; 2 day treatment period, discharge and follow-up
Population: A comparison between treatment groups was performed separately for each AUC with an ANCOVA model with AUC as dependent variable, treatment as fixed effect and baseline SA (0 hours) as covariate. The AUC is a cumulative measure, comparison could be performed only within the same time period therefore data was normalised over time.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel
Number analyzed (Participants) | 27 | 12 | 24
units on a scale
  Treatment period | 64.3 (28.9) | 54.5 (33.1) | 76.8 (35.2)
  Treatment to discharge | 159.0 (85.8) | 139.5 (98.6) | 245.8 (121.8)
  Treatment to follow-up | 964.3 (335.8) | 911.5 (380.1) | 1041.0 (414.4)
Statistical Analysis 1: Comparison: XF-73 2.0 mg/g Nasal Gel vs Placebo Nasal Gel; Test type: Superiority or Other; p = 0.028, ANCOVA — The adjusted means were compared for the two-day treatment period
Statistical Analysis 2: Comparison: XF-73 2.0 mg/g Nasal Gel vs Placebo Nasal Gel; Test type: Superiority or Other; p < 0.001, ANCOVA — The adjusted means were compared for the two-day treatment period to discharge
Statistical Analysis 3: Comparison: XF-73 0.5 mg/g Nasal Gel vs Placebo Nasal Gel; Test type: Superiority or Other; p = 0.005, ANCOVA — The adjusted means were compared for the two-day treatment period through to discharge

5. Secondary Outcome: The Number of Participants With Changes in Vital Signs, ECG and Routine Haematology, Clinical Chemistry and Urinalysis Tests.
Time Frame: Assessed over the two day treatment period and follow-up at 7 and 14 days relative to the first dose.
Measure: Number; unit: participants
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel
Number analyzed (Participants) | 27 | 12 | 24
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening, treatment days 1 and 2 and follow up on days 7 and 14.
Arm/Group | XF-73 2.0 mg/g Nasal Gel | XF-73 0.5 mg/g Nasal Gel | Placebo Nasal Gel
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/12 | 0/24
Other Adverse Events (participants affected / at risk) | 9/27 | 2/12 | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XF-73 2.0 mg/g Nasal Gel (N=27) | XF-73 0.5 mg/g Nasal Gel (N=12) | Placebo Nasal Gel (N=24)
rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other